CLINICAL TRIAL: NCT01990352
Title: A Single Arm Phase II Trial to Assess Association of BRCA1 Protein Expression With Overall Response Rate in Patients With Metastatic Breast Cancer on Pegylated Liposomal Doxorubicin
Brief Title: Correlate BRCA1 Protein Expression With Response to DNA Damaging Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI determined that study specimens being obtained did not yield sufficient data to analyze the prespecified outcome measures and decided to terminate the study prior to meeting enrollment goals.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1300000710
Record Dates: First submitted 2013-11-08; First posted 2013-11-21 (Estimated); Results first posted 2023-10-26 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegylated liposomal doxorubicin (Experimental): The enrolled patients will be treated with pegylated liposomal doxorubicin at 30mg/m2 every 21 days.
  Interventions: Drug: Pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — Doxil will be administered intravenously at 30mg/m2 on days 1 of a 21 day cycle.
  Other Names: Doxil

SUMMARY:
Primary Objective: To evaluate if low BRCA1 protein expression has a preferential effect on response when metastatic breast cancer patients are treated with DNA damaging chemotherapy agent, compared to historical controls

Secondary Objective: To evaluate if low BRCA1 protein expression has a preferential effect on tumor progression when metastatic breast cancer patients are treated with DNA damaging chemotherapy agent, compared to historical controls

DETAILED DESCRIPTION:
DNA is constantly subject to damage from exposures including drugs (including chemotherapy), sunlight and aging. Certain genes in the human body help repair this damage (i.e. BRCA1 and other genes). The purpose of this study is to find out if BRCA1 protein expression has a role in response to chemotherapy drugs.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer and have formalin-fixed, paraffin embedded primary tumor available for testing BRCA1 protein expression
* Adults over 18 years of age
* Have resolution of all acute toxic effects of any prior chemotherapy or radiotherapy to NCI CTC grade ≤ 1 prior to study registration.
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study specific screening procedures
* Be willing and able to comply with the treatment plan, scheduled clinic visits, laboratory and oncological tests and other study procedures
* Have a ECOG performance status of 0 - 2
* Measurable disease by CT by RECIST 1.1 to evaluate response
* Adequate bone marrow function defined as platelets 100 X 109 cells/L, neutrophils 1.5 x 109 cells/L, white blood cells (WBC) 3.0 x 109 cells/L and a hemoglobin 90 gm/L
* Creatinine < 1.5 mg/dl or creatinine clearance > 40 ml/min
* Liver function tests (AST and or ALT) should be 2 x upper limit of normal (ULN, defined as per laboratory where blood testing is done), total bilirubin 1.5 x ULN (except for patients with liver metastases, ALT and/or ALT 5 times the upper limit of normal is accepted)

Exclusion Criteria:

* Myocardial infarction within 6 months of registration
* Brain metastases unless documented to be controlled post completion of local therapy (surgery and/or radiation therapy) for at least four weeks prior to registration
* Pregnant or breast feeding women. Women with child bearing potential must use effective measures to prevent pregnancy while receiving pegylated liposomal doxorubicin
* Have a concurrent active non-breast malignancy except for non-melanoma skin cancer
* Her2 positive tumors as defined by FDA guidelines(3+ immunohistochemical staining, defined as uniform, intense membrane staining of more than 10% of invasive tumor cells, and for cases with 2+ staining showing gene amplification by FISH, expressed as a ratio of more than 2 when comparing HER-2 gene and chromosome 17 fluorescent signals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalisani, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegylated Liposomal Doxorubicin
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants]
  <=69 years | 18
  >=70 years | 5
  Unknown | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate for Metastatic Breast Cancer Patients With Low BRCA1 Protein Expression in Their Tumor, Treated With Pegylated Liposomal Doxorubicin
Description: Evaluating if low BRCA1 protein expression has a preferential effect on response when metastatic breast cancer patients are treated with DNA damaging chemotherapy agent, compared to historical controls. Response rate is defined as the percentage of evaluable patients who achieve complete response (CR) or partial response (PR) as measured by RECIST 1.1 on CT or PET/CT as the best overall response.
Time Frame: Start of treatment and repeat imaging done at 9 weeks (± 7 days)
Population: The assay to evaluate BRCA1 protein expression failed to assess due to a multitude of reasons. It could not be validated, and the collaborator discontinued the assay's further development. Since were were not able to perform the BRCA1 protein expression, the analysis for overall response rate was not performed and we are unable to report any data.
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival for Patients With Breast Cancer With Low BRCA1 Protein Expression Treated With Pegylated Liposomal Doxorubicin
Description: Evaluating if low BRCA1 protein expression has a preferential effect on tumor progression when metastatic breast cancer patients are treated with DNA damaging chemotherapy agent, compared to historical controls. Progression free survival will be measured as the times from the start of pegylated liposomal doxorubicin to the time the patient is first recorded as having disease progression or dies. If a patient does not progress or die while being followed via tumor assessment, progression-free survival will be censored at the time of last disease assessment. The median progression free survival will be calculated in patients with low BRCA1 protein expression and intact BRCA1 protein expression. Median progression free survival will be estimated by Kaplan-Meier methodology
Time Frame: Start of Treatment until the date of first documented progression or date of death, assessed up to an expected average of 100 weeks
Population: The assay to evaluate BRCA1 protein expression failed to assess due to a multitude of reasons. It could not be validated, and the collaborator discontinued the assay's further development. Since were were not able to perform the BRCA1 protein expression, the analysis for progression-free survival was not performed and we are unable to report any data.
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed through study completion.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed through study completion.
Arm/Group | Pegylated Liposomal Doxorubicin
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The trial was started with preliminary data on BRCA1 immunohistochemistry assay developed with a collaborator. The assay, in the trial, due to differences in the timeline on when the tumor tissue was collected, the variability in the tumor tissue processing, storage, and age of the samples, the assay did not work on the samples as projected. Subsequently, due to COVID-19 and the challenges with the assay performance, the collaborator discontinued further development of the assay.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT01990352/Prot_SAP_000.pdf